CLINICAL TRIAL: NCT02372513
Title: The Frequency of Cholesteryl Ester Storage Disease in Children With Unexplained Transaminase Elevation and Chronic Liver Disease
Brief Title: National Lysosomal Acid Lipase Deficiency Study
Acronym: LAL-D
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Zarife Kuloglu, Professor (M.D.), Ankara University
Other Study IDs: LALD-TR
Record Dates: First submitted 2015-02-21; First posted 2015-02-26 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cholesteryl Ester Storage Disease
Keywords: Cholesteryl Ester Storage Disease; Children; Liver disease
MeSH Terms: conditions — Cholesterol Ester Storage Disease; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Cholesteryl Ester Storage Disease (CESD) is an autosomal recessive lysosomal storage disorder (LSD) caused by mutations in the lysosomal acid lipase gene (LIPA) that markedly reduce lysosomal acid lipase (LAL) activity, leading to the accumulation of lipids, predominately cholesteryl esters and triglycerides, in various tissues and cell types. In the liver, accumulation of lipids leads to diffuse microvesicular steatosis, which progresses to fibrosis and ultimately, to micronodular cirrhosis. Patients typically present with hepatomegaly, liver dysfunction, hepatic failure and type II hyperlipidemia. Although hepatosteatosis is a typical finding, the liver biopsy diagnosis may be misclassified as non-alcoholic fatty liver disease, non-alcoholic steatohepatitis or cryptogenic liver disease. Biopsy and radiological findings are not considered diagnostic, but help to suspicion of CESD. The definitive diagnosis is based on deficient LAL activity and/or LIPA gene mutations.

CESD is pan-ethnic, however, the disease incidence is unknown. The estimated incidence of the disease indicates that CESD should be largely underdiagnosed especially in European patients. Elevation of serum transaminases, and hepatomegaly are early indications of liver impairment. Therefore, CESD should be considered as a differential diagnosis in liver disease of unknown origin.

To data, there is no study which evaluated the frequency of CESD in children with unexplained transaminase elevation and/or organomegaly and/or chronic liver disease. The aim of this prospective, multicenter and cross-sectional study is to investigate frequency of CESD in children with unexplained transaminase elevation and/or and/or chronic liver disease and to identify demographic and clinical features of CESD.

DETAILED DESCRIPTION:
Patients of 3 months to 18 years of age at the time of enrolment who have unexplained transaminase elevation (serum alanine aminotransferase (ALT) levels > 1.5 times the upper limit of normal) for more than 3 months and/or unexplained hepatomegaly or hepatosplenomegaly and/or obesity- unrelated hepatosteatosis and/or biopsy-proven cryptogenic fibrosis and cirrhosis and/or liver transplantation for cryptogenic cirrhosis will be included.

Potential participants will be invited for LAL enzyme analysis. Written informed consent will be obtained from the parents or guardians of the participants at the time of enrolment. Prospective and retrospective data will be collected. Complete family and medical history, physical examination and previously existing laboratory findings will be recorded on standard case reports form and up to 0.25 ml of blood will be drawn for LAL enzyme analysis. The blood obtained from participants will be spotted on filter paper, and dried blood spot sample (DBS) will be prepared. Finally, the dried blood spot sample will be sent to reference laboratory (NHS Greater Glasgow and Clyde, England) for LAL enzyme measurement within 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female of 3 months to 18 years of age at the time of enrolment
2. Patients who have unexplained transaminase elevation (serum ALT levels > 1.5 times the upper limit of normal) for more than 3 months
3. Patients who have unexplained hepatomegaly or hepatosplenomegaly
4. Patients who have obesity- unrelated hepatosteatosis
5. Patients who have biopsy-proven cryptogenic fibrosis and cirrhosis
6. Patients with liver transplantation for cryptogenic cirrhosis

Exclusion Criteria:

1. A male or female < 3 months or > 18 years old
2. Patients with obesity -related hepatosteatosis
3. Patients with drug-induced hepatosteatosis ( such as aspirin, methotrexate, amiodarone, glucocorticoid, tamoxifen, 5-fluorouracil, valproate, nucleoid revers transcriptase inhibitors)
4. Patients with organomegaly or transaminase elevation due to infectious causes (EBV, Brucella, cytomegalovirus, salmonella, malaria, leishmania etc), hæmato-oncological disease (hemolytic anemia, leukemia,lymphoma, malign or benign liver neoplasms), connective tissue disorders (SLE, RA), cardiac and vascular causes (heart failure, pericarditis, Budd-Chiari syndrome, portal vein thrombosis) and obesity.
5. Patient with definitive diagnosed chronic liver disease such as chronic viral hepatitis (B, C hepatitis), autoimmune hepatitis, alpha-1 antitrypsin deficiency, Wilson disease, metabolic disorders.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients of 3 months to 18 years of age at the time of enrolment who have unexplained transaminase elevation (serum ALT levels > 1.5 times the upper limit of normal) for more than 3 months and/or unexplained hepatomegaly or hepatosplenomegaly and/or obesity- unrelated hepatosteatosis and/or biopsy-proven cryptogenic fibrosis and cirrhosis and/or liver transplantation for cryptogenic cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01-31 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Frequency of Cholesteryl Ester Storage Disease in children who have unexplained transaminase elevation for more than 3 months and/or organomegaly and/or hepatosteatosis unrelated to obesity and/or cryptogenic fibrosis and cirrhosis | First day

SECONDARY OUTCOMES:
Identify demographic and clinical features of Cholesteryl Ester Storage Disease | First day

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Kuloglu, M.D, Study Director — Ankara University
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Reynolds T. Cholesteryl ester storage disease: a rare and possibly treatable cause of premature vascular disease and cirrhosis. J Clin Pathol. 2013 Nov;66(11):918-23. doi: 10.1136/jclinpath-2012-201302. Epub 2013 Sep 2. PMID 23999269
- [Background] Hulkova H, Elleder M. Distinctive histopathological features that support a diagnosis of cholesterol ester storage disease in liver biopsy specimens. Histopathology. 2012 Jun;60(7):1107-13. doi: 10.1111/j.1365-2559.2011.04164.x. PMID 22621222
- [Background] Zhang B, Porto AF. Cholesteryl ester storage disease: protean presentations of lysosomal acid lipase deficiency. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):682-5. doi: 10.1097/MPG.0b013e31828b36ac. PMID 23403440
- [Background] Hamilton J, Jones I, Srivastava R, Galloway P. A new method for the measurement of lysosomal acid lipase in dried blood spots using the inhibitor Lalistat 2. Clin Chim Acta. 2012 Aug 16;413(15-16):1207-10. doi: 10.1016/j.cca.2012.03.019. Epub 2012 Mar 29. PMID 22483793
- [Background] Dairaku T, Iwamoto T, Nishimura M, Endo M, Ohashi T, Eto Y. A practical fluorometric assay method to measure lysosomal acid lipase activity in dried blood spots for the screening of cholesteryl ester storage disease and Wolman disease. Mol Genet Metab. 2014 Feb;111(2):193-6. doi: 10.1016/j.ymgme.2013.11.003. Epub 2013 Nov 16. PMID 24295952
- [Background] Ambler GK, Hoare M, Brais R, Shaw A, Butler A, Flynn P, Deegan P, Griffiths WJ. Orthotopic liver transplantation in an adult with cholesterol ester storage disease. JIMD Rep. 2013;8:41-6. doi: 10.1007/8904_2012_155. Epub 2012 Jul 24. PMID 23430518
- [Background] Dalgic B, Sari S, Gunduz M, Ezgu F, Tumer L, Hasanoglu A, Akyol G. Cholesteryl ester storage disease in a young child presenting as isolated hepatomegaly treated with simvastatin. Turk J Pediatr. 2006 Apr-Jun;48(2):148-51. PMID 16848116
- [Background] Balwani M, Breen C, Enns GM, Deegan PB, Honzik T, Jones S, Kane JP, Malinova V, Sharma R, Stock EO, Valayannopoulos V, Wraith JE, Burg J, Eckert S, Schneider E, Quinn AG. Clinical effect and safety profile of recombinant human lysosomal acid lipase in patients with cholesteryl ester storage disease. Hepatology. 2013 Sep;58(3):950-7. doi: 10.1002/hep.26289. Epub 2013 Mar 28. PMID 23348766
- [Result] Bernstein DL, Hulkova H, Bialer MG, Desnick RJ. Cholesteryl ester storage disease: review of the findings in 135 reported patients with an underdiagnosed disease. J Hepatol. 2013 Jun;58(6):1230-43. doi: 10.1016/j.jhep.2013.02.014. Epub 2013 Feb 26. PMID 23485521
- [Result] Fasano T, Pisciotta L, Bocchi L, Guardamagna O, Assandro P, Rabacchi C, Zanoni P, Filocamo M, Bertolini S, Calandra S. Lysosomal lipase deficiency: molecular characterization of eleven patients with Wolman or cholesteryl ester storage disease. Mol Genet Metab. 2012 Mar;105(3):450-6. doi: 10.1016/j.ymgme.2011.12.008. Epub 2011 Dec 17. PMID 22227072
- [Result] Fouchier SW, Defesche JC. Lysosomal acid lipase A and the hypercholesterolaemic phenotype. Curr Opin Lipidol. 2013 Aug;24(4):332-8. doi: 10.1097/MOL.0b013e328361f6c6. PMID 23652569
- [Result] Reiner Z, Guardamagna O, Nair D, Soran H, Hovingh K, Bertolini S, Jones S, Coric M, Calandra S, Hamilton J, Eagleton T, Ros E. Lysosomal acid lipase deficiency--an under-recognized cause of dyslipidaemia and liver dysfunction. Atherosclerosis. 2014 Jul;235(1):21-30. doi: 10.1016/j.atherosclerosis.2014.04.003. Epub 2014 Apr 15. PMID 24792990
- [Result] Muntoni S, Wiebusch H, Jansen-Rust M, Rust S, Seedorf U, Schulte H, Berger K, Funke H, Assmann G. Prevalence of cholesteryl ester storage disease. Arterioscler Thromb Vasc Biol. 2007 Aug;27(8):1866-8. doi: 10.1161/ATVBAHA.107.146639. No abstract available. PMID 17634524
- [Result] Scott SA, Liu B, Nazarenko I, Martis S, Kozlitina J, Yang Y, Ramirez C, Kasai Y, Hyatt T, Peter I, Desnick RJ. Frequency of the cholesteryl ester storage disease common LIPA E8SJM mutation (c.894G>A) in various racial and ethnic groups. Hepatology. 2013 Sep;58(3):958-65. doi: 10.1002/hep.26327. Epub 2013 Jul 29. PMID 23424026